CLINICAL TRIAL: NCT05507541
Title: Phase 2 Study With Safety run-in of PD-1 Inhibitor and IgG4 SIRPα-Fc Fusion Protein (TTI-622) in Relapsed Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: TTI-622 in Combination With Pembrolizumab for the Treatment of Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC200802; NCI-2022-06277 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-003869 (Registry Identifier: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Recurrent ALK Positive Large B-Cell Lymphoma; Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Diffuse Large B-Cell Lymphoma Associated With Chronic Inflammation; Recurrent Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent EBV-Positive Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Recurrent Grade 3b Follicular Lymphoma; Recurrent High Grade B-Cell Lymphoma; Recurrent High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Recurrent High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Recurrent High Grade B-Cell Lymphoma, Not Otherwise Specified; Recurrent Intravascular Large B-Cell Lymphoma; Recurrent Primary Cutaneous Diffuse Large B-Cell Lymphoma, Leg Type; Recurrent Primary Mediastinal (Thymic) Large B-Cell Lymphoma; Recurrent T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Refractory ALK Positive Large B-Cell Lymphoma; Refractory Diffuse Large B-Cell Lymphoma Associated With Chronic Inflammation; Refractory Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory EBV-Positive Diffuse Large B-Cell Lymphoma, Not Otherwise Specified; Refractory Grade 3b Follicular Lymphoma; Refractory High Grade B-Cell Lymphoma; Refractory High Grade B-Cell Lymphoma With MYC and BCL2 or BCL6 Rearrangements; Refractory High Grade B-Cell Lymphoma With MYC, BCL2, and BCL6 Rearrangements; Refractory High Grade B-Cell Lymphoma, Not Otherwise Specified; Refractory Intravascular Large B-Cell Lymphoma; Refractory Primary Cutaneous Diffuse Large B-Cell Lymphoma, Leg Type; Refractory Primary Mediastinal Large B-Cell Lymphoma; Refractory T-Cell/Histiocyte-Rich Large B-Cell Lymphoma; Recurrent Gray Zone Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — Specimen Handling; TTI-621; pembrolizumab; Magnetic Resonance Spectroscopy; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (pembrolizumab, TTI-621) -- CLOSED TO ACCRUAL 8/16/2024 (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle and TTI-621 IV over 60-120 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT scans or CT scans of the chest, abdomen, and pelvis prior to cycle 3 and every 4 cycles thereafter. If no disease progression after cycle 12, patients then receive pembrolizumab IV over 30 minutes on day 1 of each cycle and TTI-621 IV over 60 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 23 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT and/or CT and blood sample collection throughout the study. Patients may undergo biopsy on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Ontorpacept; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Procedure: Biopsy
- Arm B (pembrolizumab, TTI-622) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle and TTI-622 IV over 60-90 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT scans or CT scans of the chest, abdomen, and pelvis prior to cycle 3 and every 4 cycles thereafter. If no disease progression after cycle 12, patients then receive pembrolizumab IV over 30 minutes on days 1 of each cycle and TTI-622 IV over 60-90 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 23 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Drug: Maplirpacept; Procedure: Biopsy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection; Blood Sample Collection
Procedure: Computed Tomography — Undergo PET/CT or CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography; Computerized axial tomography (procedure)
Drug: Ontorpacept — Given IV
  Other Names: SIRPa-Fc Fusion Protein TTI-621; SIRPaFc; TTI 621; TTI-621
  Arms: Arm A (pembrolizumab, TTI-621) -- CLOSED TO ACCRUAL 8/16/2024
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Procedure: Positron Emission Tomography — Undergo PET/CT scans
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; Positron emission tomography (procedure)
Drug: Maplirpacept — Given IV
  Other Names: SIRPa-IgG4 Fc; SIRPa-IgG4 Fc TTI-622; TTI 622; TTI-622; TTI622; SIRPa-IgG4-Fc Fusion Protein TTI-622
  Arms: Arm B (pembrolizumab, TTI-622)
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx

SUMMARY:
This phase II trial tests the safety, side effects, and best dose of TTI-621 (closed to enrollment) or TTI-622 in combination with pembrolizumab in treating patients with diffuse large B-cell lymphoma that has come back after a period of improvement (relapsed) or that does not respond to treatment (refractory). TTI-621 and TTI-622 are called fusion proteins. A fusion protein includes two specialized proteins that are joined together. In TTI-621 and TTI-622, one of the proteins binds with other proteins found on the surface of certain cells that are part of the immune system. The other protein targets and blocks a protein called CD47. CD47 is present on cancer cells and is used by those cells to hide from the body's immune system. By blocking CD47, TTI-621 and TTI-622 may help the immune system find and destroy cancer cells. Pembrolizumab is a monoclonal antibody directed against human cell surface receptor PD-1 (programmed death-1 or programmed cell death-1) that works by helping the body's immune system attack the cancer and may interfere with the ability of cancer cells to grow and spread. Giving TTI-621 (closed to enrollment) or TTI-622 in combination with pembrolizumab may kill more cancer cells in patients with relapsed or refractory diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the toxicities of maplirpacept (TTI-622) combined with pembrolizumab and to identify the recommended phase 2 dose (RP2D) of TTI-622, combined with pembrolizumab. (Safety run-in) II. To estimate preliminary efficacy of pembrolizumab in combination with TTI-622 as measured by overall response rate (ORR). (Phase 2).

SECONDARY OBJECTIVE:

I. To estimate efficacy of pembrolizumab in combination with TTI-622 as measured by duration of response (DOR), progression free survival (PFS), and overall survival (OS).

CORRELATIVE OBJECTIVE:

I. Correlation of biomarkers measured in serial peripheral blood samples and tumor tissues with clinical responses, which may include but are not limited to: SIRPalpha expression, monocyte/macrophage markers in tumor micro-environment, tumor infiltrating lymphocytes (TILs), PD-1/PDL-1 expression.

OUTLINE: Patients are assigned to 1 of 2 arms. Patients enrolling after 8/16/2024 are assigned to Arm B.

ARM A (CLOSED TO ACCRUAL AS OF 8/16/2024): Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle and ontorpacept (TTI-621) IV over 60-120 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo positron emission tomography/computed tomography (PET/CT) scans or CT scans of the chest, abdomen, and pelvis prior to cycle 3 and every 4 cycles thereafter. If no disease progression after cycle 12, patients then receive pembrolizumab IV over 30 minutes on day 1 of each cycle and TTI-621 IV over 60 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 23 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT and/or CT and blood sample collection throughout the study. Patients may undergo biopsy on study.

ARM B: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle and TTI-622 IV over 60-90 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT scans or CT scans of the chest, abdomen, and pelvis prior to cycle 3 and every 4 cycles thereafter. If no disease progression after cycle 12, patients then receive pembrolizumab IV over 30 minutes on day 1 of each cycle and TTI-622 IV over 60-90 minutes on day 1 of each cycle. Treatment repeats every 21 days for up to 23 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo PET/CT and/or CT and blood sample collection throughout the study. Patients may undergo biopsy on study.

After completion of the study treatment, patients are followed every 6 months for up to 2 years from registration.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Documented CD20+ mature B-cell neoplasm according to World Health Organization (WHO) classification (Swerdlow et al., 2016) as one of the following:

  * Diffuse large B-cell lymphoma not otherwise specified (NOS) including

    * Transformed lymphoma
    * Richter's transformation
    * Germinal center B-cell type
    * Activated B-cell type
  * High-grade B-cell lymphoma (HGBCL), NOS
  * Primary mediastinal (thymic) large B-cell lymphoma
  * Patients with "double-hit" or "triple-hit" diffuse large B-cell lymphoma (DLBCL) (technically as HGBCL, with MYC and BCL2 and/or BCL6 rearrangements)
  * Follicular lymphoma 3B
  * T-cell/histiocyte-rich large B cell lymphoma
  * Large B-cell lymphoma with IRF4 rearrangement
  * Primary cutaneous DLBCL, leg type
  * Epstein-Barr virus (EBV) positive DLBCL, NOS
  * DLBCL associated with chronic inflammation
  * Intravascular large B-cell lymphoma
  * ALK positive large B-cell lymphoma
* Relapsed, progressive and/or refractory disease (Cheson et al., 2007) following treatment with an anti-CD20 monoclonal antibody (e.g., rituximab) in combination with chemotherapy
* Measurable disease as defined below:

  * Fluorodeoxyglucose (FDG)-avid lymphomas: Measurable disease with computerized tomography (CT) (or magnetic resonance imaging [MRI]) scan with involvement of 2 or more clearly demarcated lesions/nodes with a long axis > 1.5 cm and short axis > 1.0 cm (or 1 clearly demarcated lesion/node with a long axis > 2.0 cm and short axis >= 1.0 cm) AND FDG positron emission tomography (PET) scan that demonstrates positive lesion(s) compatible with CT (or MRI) defined anatomical tumor sites
  * FDG-nonavid lymphomas: Measurable disease with CT (or MRI) scan with involvement of 2 or more clearly demarcated lesions/nodes with a long axis > 1.5 cm and short axis > 1.0 cm or 1 clearly demarcated lesion/node with a long axis > 2.0 cm and short axis >= 1.0 cm.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* >= 4 weeks from last dose of anti-CD20 targeting therapy
* >= 12 weeks post chimeric antigen receptor (CAR) T-cell therapy
* Resolution of all adverse events due to prior therapy to =< Grade 1 or baseline NOTE: Patients with =< Grade 2 neuropathy may be eligible. Patients with endocrine-related adverse events (AEs) Grade =< 2 requiring treatment or hormone replacement may be eligible
* If receiving glucocorticoid treatment at screening, treatment must be tapered down and administered with a maximum of 10 mg daily in the last 14 days prior to registration
* Absolute neutrophil count (ANC) >= 500/mm^3; growth factor support allowed in case of bone marrow involvement (obtained =< 7 days prior to registration)
* Absolute lymphocyte count >= 200/mm^3 (obtained =< 7 days prior to registration)
* Platelet count >= 75,000/mm^3 (obtained =< 7 days prior to registration)
* Hemoglobin >= 8.0 g/dL (obtained =< 7 days prior to registration)
* International normalized ratio (INR) or activated partial thromboplastin time (aPTT) =< 1.5 × upper limit of normal (ULN) unless participant is receiving anticoagulant therapy as long as prothrombin time (PT) or aPTT is within therapeutic range of intended use of anticoagulants (obtained =< 7 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN), unless due to Gilbert's disease (direct bilirubin [bili] =< ULN) (obtained =< 7 days prior to registration)
* Aspartate transaminase [AST/serum glutamic oxaloacetic transaminase (SGOT)] and alanine transaminase [ALT/serum glutamic pyruvic transaminase (SGPT)] =< 2.5 x ULN (obtained =< 7 days prior to registration)
* Calculated creatinine clearance >=30 mL/min using the Cockcroft-Gault formula (obtained =< 7 days prior to registration)
* Provide informed written consent
* Negative pregnancy test done =< 3 days prior to registration, for persons of childbearing potential only
* Female of childbearing must agree to use a highly effective method of contraception during the treatment and for 120 days after the last dose of study treatment
* Male participants with female partners of childbearing potential must agree to refrain from donating sperm and one of the conception methods during the treatment and for 120 days after last dose study treatment
* Willing to return to the enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing to provide mandatory tissue and blood samples for correlative research purposes

Exclusion Criteria:

* Primary central nervous system (CNS) lymphoma or known CNS involvement by lymphoma at screening as confirmed by magnetic resonance imaging (MRI)/computed tomography (CT) scan (brain) and, if clinically indicated, by lumbar puncture
* Known past or current malignancy other than inclusion diagnosis, except for:

  * Cervical carcinoma of Stage 1B or less
  * Non-invasive basal cell or squamous cell skin carcinoma
  * Non-invasive, superficial bladder cancer
  * Prostate cancer with a current prostate specific antigen (PSA) level < 0.1 ng/mL
  * Any curable cancer with a complete response (CR) of > 2 years duration
* Received < 2 prior systemic anti-cancer therapy including investigational agents =< 4 weeks or =< 5 half-lives, whichever is shorter, prior to registration
* Received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX-40, CD137) =< 4 weeks prior to registration
* Known clinically significant cardiac disease, including:

  * Onset of unstable angina pectoris within 6 months of signing informed consent form (ICF)
  * Acute myocardial infarction within 6 months of signing ICF
  * Congestive heart failure (grade III or IV as classified by the New York Heart Association and/or known decrease ejection fraction of < 45%)
* Chronic ongoing infectious diseases (except hepatitis B or hepatitis C) requiring treatment (excluding prophylactic treatment) at the time of enrollment or =< the previous 2 weeks
* Confirmed history or current autoimmune disease or other diseases resulting in permanent immunosuppression or requiring permanent immunosuppressive therapy or primary immunodeficiency disorder. Low-dose steroids (=< 10 mg daily of prednisone equivalent) is allowed
* Seizure disorder requiring therapy (such as steroids or anti-epileptics)
* Autologous hematopoietic stem cell transplant (HSCT) =< 100 days prior or any prior allogeneic HSCT or solid organ transplantation
* Known human immunodeficiency virus (HIV) infection
* Exposed to live or live attenuated vaccine =< 4 weeks prior to registration
* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons
  * Nursing persons
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Patient has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the patient (e.g., compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to:

  * ongoing or active infection
  * uncontrolled infection requiring ongoing antibiotics

    * symptomatic congestive heart failure
    * unstable angina pectoris
    * cardiac arrhythmia
    * or psychiatric illness/social situations that would limit compliance with study requirements
    * known substance abuse disorder
* Known hypersensitivity to pembrolizumab
* Major surgery other than diagnostic surgery =< 4 weeks prior to registration
* Prior radiation therapy =< 2 weeks prior to registration or who has not recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. Note: A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-CNS disease
* Active autoimmune disease such as Crohn's disease, rheumatoid arthritis, Sjogren's disease, systemic lupus erythematosus, or similar conditions requiring systemic treatment =< the past 3 months or a documented history of clinically severe autoimmune disease/syndrome difficult to control in the past.

EXCEPTIONS:

* Vitiligo or resolved childhood asthma/atopy
* Intermittent use of bronchodilators or local steroid injections
* Hypothyroidism stable on hormone replacement,
* Diabetes stable with current management
* History of positive Coombs test but no evidence of hemolysis
* Psoriasis not requiring systemic treatment
* Conditions not expected to recur in the absence of an external trigger

  * Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (HCV) (defined as HCV ribonucleic acid [RNA] is detected) infection
  * Prior anti CD47 therapy
  * Active use of anticoagulant like warfarin. Use of low molecular weight heparin and factor Xa inhibitors will be permitted on case by case basis. There will be no restriction for daily aspirin < 81mg daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose of maplirpacept (TTI-622) when given in combination with pembrolizumab (Safety run-in) | Up to 6 weeks
  Defined as the highest dose for which at most 1 out of 6 subjects experience significant toxicity during the 6-week safety assessment period. Toxicity will be measured per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5. Significant toxicity is defined as an adverse event occurring during the first cycle of treatment that is possibly, probably, or definitely related to study treatment.
Overall response (Phase 2) | Up to 2 years
  A success is defined as an objective status of partial metabolic response (PMR) or complete metabolic response (CMR) by positron emission tomography-computed tomography (PET-CT) based criteria at any time. The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Note: For patients where PET/CT scan was not available due to insurance coverage and who received a CT scan only, they will still be considered evaluable for the primary endpoint and will be included in the denominator for estimating overall response rate. In these patients, the CT-based responses will be reported descriptively.

SECONDARY OUTCOMES:
Duration of response (DOR) (Phase 2) | Up to 2 years
  Defined for all evaluable patients who have achieved an objective response as the date at which the patient's objective status is first noted to be either a CMR or PMR to first documentation of disease progression. DOR will be descriptively summarized.
Incidence of adverse events (AEs) (Phase 2) | Up to 2 years
  All eligible patients that have initiated treatment will be considered evaluable for assessing AE rate(s). The maximum grade for each type of AE will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the AE(s) to the study treatment will be taken into consideration.
Overall survival (OS) (Phase 2) | up to 2 years
  OS is defined as the time from registration to death due to any cause.
Progression-free survival (PFS) (Phase 2) | Up to 2 years
  PFS is defined as the time from registration to the first documentation of disease progression [progressive metabolic disease (PMD) or progressive disease (PD)] or death due to any cause in the absence of documented progression.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M. Ansell, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials